CLINICAL TRIAL: NCT06649110
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of LTP001 in Healthy Adult Participants (Part A) and to Evaluate the Efficacy and Safety of LTP001 for the Treatment of Participants With Pulmonary Arterial Hypertension (Part B)
Brief Title: A Study to Learn About the Treatment LTP001 in Healthy Participants (Part A) and in Participants With PAH (Part B)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLTP001A12202
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers, Pulmonary Arterial Hypertension
Keywords: LTP001; pulmonary arterial hypertension; PAH; PVR
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LTP001 Dose 1 (Experimental)
  Interventions: Drug: LTP
- LTP001 Dose 2 (Experimental)
  Interventions: Drug: LTP
- LTP001 Dose 3 (Experimental)
  Interventions: Drug: LTP
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LTP — LTP001
  Arms: LTP001 Dose 1; LTP001 Dose 2; LTP001 Dose 3
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A study to learn about the treatment LTP001 in healthy participants (Part A) and in participants with PAH (Part B)

DETAILED DESCRIPTION:
The CLTP001A12202 study will explore the safety, tolerability, and pharmacokinetics of LTP001 in healthy volunteers (Part A) and will evaluate the safety and efficacy (Part B) followed by safety extension in participants with pulmonary arterial hypertension.

ELIGIBILITY:
Part A Inclusion Criteria:

* Healthy males and non-child-bearing potential females

Part A Exclusion Criteria:

* Clinically significant ECG or cardiac abnormalities, any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the participant in the study Other protocol-defined inclusion/exclusion criteria may apply.
* For Japanese cohorts: participants per protocol should be first generation Japanese or up to third generation Japanese as defined in inclusion criteria 7 of the protocol.

Part B Inclusion Criteria:

-Confirmed diagnosis of PAH, pre-randomization PVR ≥400 dyn.sec.cm-5, treatment with stable doses of standard-of-care PAH therapies, 6-minute walk distance ≥ 150 m and ≤450 m.

Part B Exclusion Criteria:

Any surgical or medical condition which may place the participant at higher risk from his/her participation in the study Women of child-bearing potential unless they are using highly effective methods of contraception Sexually active males unwilling to use a condom during intercourse while taking study treatment and for 24 hours after stopping study treatment.

History of hypersensitivity to any of the study treatments or excipients

Other protocol-defined inclusion / exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2028-11-29 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Part A- Number of participants with Adverse events (AEs) and Serious Adverse events (SAEs) | Baseline to Day 35
  Safety endpoints, including vital signs, ECG, clinical laboratory evaluations and adverse events up to and including the end-of-study visit.
Part B-Treatment Period 1: Change in pulmonary vascular resistance (PVR) | Baseline to Week 24
  PVR is a hemodynamic variable of pulmonary circulation and is measured by right heart catheterization.
Part B-Treatment Period 2: Number of participants with Adverse events (AEs) and Serious Adverse events (SAEs) | From Day 1 until Week 106
  Safety endpoints, including vital signs, ECG, clinical laboratory evaluations, treatment-emergent adverse events and discontinuations due to adverse events.

SECONDARY OUTCOMES:
Part A- Maximum observed plasma concentrations (Cmax) | Baseline to Day 35
  Cmax is defined as the maximum (peak) observed concentration following a dose.
Part A- Time to reach maximum plasma concentration (Tmax) | Baseline to Day 35
  Tmax is defined as the time to reach maximum (peak) concentration following a dose.
Part A- Area under plasma concentration-time curve from time zero to the last measurable concentration sampling time (AUClast) | Baseline to Day 35
  AUClast is the area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (tlast).
Part A- Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC[0-inf]) | Baseline to Day 35
  The AUC is the area under the plasma concentration from time zero to infinity (mass x time x volume-1).
Part A- Terminal elimination half-life (T1/2) | Baseline to Day 35
  T1/2 is the elimination half-life associated with the terminal slope.
Part B-Treatment Period 1: Change in the Six-minute Walk Test (6MWT) | Baseline to Week 24
  The 6MWD test is self-paced, with standardized instructions and encouragement being given as participants walk as far as possible over 6 minutes through a flat corridor.
Part B-Treatment Period 1: Change in N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline to Week 24
  N-terminal pro brain natriuretic peptide (NTproBNP) are peptide (small proteins) that are either hormones or part of the peptide that contained the hormone at one time. They are continually produced in small quantities in the heart and released in larger quantities when the heart senses that it needs to work harder, as in heart failure.
Part B-Treatment Period 1: Change in World Health Organization (WHO) functional class (FC) | Baseline to Week 24
  The Investigator or study staff will assign a WHO functional class to a participant based on reports of symptoms and activity limitation.
  * Class I: symptom-free when physically active or resting.
  * Class II: no symptoms at rest, but normal activities such as climbing the stairs, grocery shopping, or making the bed cause some discomfort and shortness of breath.
  * Class III: resting may be symptom-free, but normal chores around the house are greatly limited due to shortness of breath and feeling tired.
  * Class IV: symptoms at rest and severe symptoms with an activity
Part B-Treatment Period 2: Change in the Six-minute Walk Test (6MWT) | Baseline to Month 18
  The 6MWD test is self-paced, with standardized instructions and encouragement being given as participants walk as far as possible over 6 minutes through a flat corridor.
Part B-Treatment Period 2: Change in World Health Organization (WHO) functional class (FC) | Baseline to Month 18
  The Investigator or study staff will assign a WHO functional class to a participant based on reports of symptoms and activity limitation.
  * Class I: symptom-free when physically active or resting.
  * Class II: no symptoms at rest, but normal activities such as climbing the stairs, grocery shopping, or making the bed cause some discomfort and shortness of breath.
  * Class III: resting may be symptom-free, but normal chores around the house are greatly limited due to shortness of breath and feeling tired.
  * Class IV: symptoms at rest and severe symptoms with an activity

CONTACTS AND LOCATIONS:
Locations (16):
- United States (7):
  - Stanford Medical Center, Stanford, California
  - U of Kansas Medical Center, Kansas City, Kansas
  - Norton Infectious Diseases Specialists, Louisville, Kentucky
  - Summit Health Eastside Clinic, Bend, Oregon
  - PPD Development LP, Austin, Texas
  - The University of Utah, Salt Lake City, Utah
  - Pul Ass Richmond Inc P A R, Richmond, Virginia
- Australia (3):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, New Lambton Heights, New South Wales
- Italy (2):
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Ivrea, TO
- Novartis Investigative Site, Riga, Latvia
- Novartis Investigative Site, Lisbon, Portugal
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Novartis.aspx